CLINICAL TRIAL: NCT07178925
Title: Follow-up Cohort of Patients With Antiphospholipid Syndrome
Acronym: ReLaps
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/353/OB; 2018-A02845-50 (Other: ANSM)
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Antiphospholipid Syndrome (APS)
Keywords: thrombotic recurrence rate; risk factors; treatment tolerance
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — A collection of biological samples will be created during this research protocol to enable the subsequent identification of endothelial, oxidative stress and coagulation parameters in these patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study of Antiphospholipid Syndrome responding to the Sydney classification of 2006 — The main objective of the research is to define the thrombotic recurrence rate in our cohort of patients followed for APS in the internal medicine department, to evaluate the complication rate associated with treatment, to search for risk factors associated with thrombotic recurrence and to define the mortality and morbidity rates of this patient population.

SUMMARY:
Antiphospholipid syndrome (APLS) is a rare pathology characterized by the association of thrombotic (arterial, venous) or obstetric clinical manifestations and the persistent presence at least twelve weeks apart of antiphospholipid antibodies (APL). It is also accompanied by accelerated atherosclerosis responsible for an increased incidence of myocardial infarction, peripheral arterial disease and stroke explaining the high cardiovascular morbidity and mortality of these patients. APS can be isolated (primary) or integrated into an autoimmune pathology such as systemic lupus erythematosus (SLE), thus defining secondary APS. Current treatment is based on anticoagulation. Currently, epidemiological data that have evaluated recurrences have estimated a rate of 5% per year. However, these studies are old and due to the significant heterogeneity of patients included in this registry, it seems that these figures are not in agreement with clinical reality.

Furthermore, several new therapeutic developments have emerged in the field of anticoagulation with the marketing of DOACs, making the EUROPHOSPHOLIPIDE data questionable. Currently, there are no clinical studies to justify the use of DOACs in this indication, but several patients have received these drugs due to intolerance or refusal of vitamin K antagonists. The other therapeutic innovation compared to the data from the EUROPHOSPHOLIPIDE cohort is the increasing use of hydroxychloroquine in clinical practice in patients with primary APS. A trial (APLAQUINE) is currently underway in our department which aims to study the endothelial protective effect of this treatment in patients with primary APS.

DETAILED DESCRIPTION:
This trial is a retrospective and prospective cohort epidemiological study whose primary objective is to determine the rate of thrombotic recurrence in our center. Secondary objectives are to determine the risk factors associated with recurrence, assess the safety of long-term treatment in this population, and evaluate the overall morbidity and mortality of this rare disease.

A better understanding of thrombotic recurrence is essential to calculate realistic population sizes for future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age and under 75 years of age
* Antiphospholipid syndrome meeting the 2006 Sydney classification

Exclusion Criteria:

* Patients under the age of 75 or over
* Syndrome not meeting the 2006 Sydney classification

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients monitored for Antiphospholipid Syndrome (APLS) in the internal medicine department
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2031-10-16 (Estimated)

PRIMARY OUTCOMES:
Thrombotic recurrence rate | Patients will be followed up in consultation every 3 months, 6 months to 1 year, for 5 years, depending on the situation. Follow-ups will not be modified compared to the usual management of the disease.
  The main objective of the research is to define the thrombotic recurrence rate in our cohort of patients followed for APS in the internal medicine department.

SECONDARY OUTCOMES:
Complication rate | Patients will be followed up in consultation every 3 months, 6 months to 1 year, for 5 years, depending on the situation. Follow-ups will not be modified compared to the usual management of the disease.
  Evaluate the complication rate associated with treatment
Risk factors associated | Patients will be followed up in consultation every 3 months, 6 months to 1 year, for 5 years, depending on the situation. Follow-ups will not be modified compared to the usual management of the disease.
  Look for risk factors associated with thrombotic recurrence
Mortality rates | Patients will be followed up in consultation every 3 months, 6 months to 1 year, for 5 years, depending on the situation. Follow-ups will not be modified compared to the usual management of the disease.
  Evaluate the mortality rates of this patient population
Morbidity rates | Patients will be followed up in consultation every 3 months, 6 months to 1 year, for 5 years, depending on the situation. Follow-ups will not be modified compared to the usual management of the disease.
  Evaluate the morbidity rates of this patient population

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.